CLINICAL TRIAL: NCT06923046
Title: Implementation of Team Clinic for Type 2 Diabetes (TCT2): A Randomized Standard Care-controlled Two-site 80-subject Clinical Trial of Shared Medical Appointment Model for Adolescents With Type 2 Diabetes
Brief Title: Implementation of Team Clinic for Type 2 Diabetes (TCT2)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: University of California, San Francisco (Other); American Diabetes Association (Other)
Responsible Party: Principal Investigator, lily chao, Principal Investigator, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CHLA-25-00070
Record Dates: First submitted 2025-03-25; First posted 2025-04-11 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care; Shared Medical Appointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Placebo Comparator): Multidisciplinary team based care every 3 months.
  Interventions: Other: Standard of Care
- Shared Medical Appointment (Active Comparator): Participants will attend 4 quarterly appointments. In addition to time with their clinician, they will also have group activities that address relevant topics.
  Interventions: Behavioral: Shared Medical Appointments

INTERVENTIONS:
Other: Standard of Care — Multidisciplinary team based care every 3 months.
  Arms: Standard Care
Behavioral: Shared Medical Appointments — Participants will attend 4 quarterly appointments. In additionto time with their clinician, they will also have groupactivities that address relevant topics.
  Arms: Shared Medical Appointment

SUMMARY:
The goal of this clinical trial is to learn if shared medical appointment is an acceptable way to deliver care to youth with type 2 diabetes.

The main question[s] it aims to answer are:

* Is shared medical appointments an acceptable care delivery model for this population?
* Does shared medical appointment improve psychosocial outcomes for this population?

Participants will attend quarterly clinic appointments and group activities and take surveys. Researchers will compare this intervention to standard of care.

ELIGIBILITY:
Patient/AYA Participants

Inclusion Criteria:

* Receives care for type 2 diabetes at either CHLA or UCSF
* English speaking youth
* Youth prescribed medication for type 2 diabetes
* English or Spanish speaking caregivers
* Age 12 to 18 years old at the time of enrollment
* Willingness to attend clinic visits and participate in group session (if randomized to Team Clinic), complete surveys

Exclusion Criteria:

* Participants who are non-verbal or unable to participate in group activities and discussions
* Pregnancy
* Inability or unwillingness of individual or legal guardian/representative to give written informed assent/consent

Caregiver/Parents Participants

Inclusion Criteria:

* Has a child between the ages of 12 and up to 18 at the time of enrollment who receives care for T2D in the endocrinology clinic at CHLA. The child must provide consent/assent to participate as a youth participant.
* Speaks English of Spanish. Over 95% of our T2D population speaks one of those two languages. Our facilitator will be bilingual in English and Spanish. It is not feasible for the facilitator to also speak another language. Having a language interpreter for discussion groups will affect the dynamics and flow of the group session
* Willingness to participate in group session (if their child is randomized to Team Clinic) and complete surveys.

Exclusion Criteria:

-Inability or unwillingness of individual to give written informed consent

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Average number of clinics attended over 1 year period to be recorded by Study Coordinator | 1 year
  Data collected is the number of patient visits to the clinic.
Change in HbA1c for patients from baseline to end of study | 1 year
  Patients' glycemic outcomes will be taken every session (Visit 0 (baseline) - Visit 4) over a one-year period
Clinic Satisfaction | 1 year
  Patient participants will complete satisfaction survey at the end of each visit using a 5-point Likert scale; "Strongly disagree" is 1, "disagree" is 2, "neutral" is 3, "agree" is 4, "strongly agree" is 5.

SECONDARY OUTCOMES:
Depression score | 1 year
  The patient health questionnaire-8 is a measure of depression severity that will be administered at baseline and again at the end of the study.
Mean time-in-range from blinded 14-day continuous glucose monitoring (CGM) for Patients between baseline and 1 year | 1 year
  A blinded CGM device will be applied to patients at enrollment and at the final study visit to capture glycemic control
Diabetes distress for patients over 1 year period | 1 year
  The Diabetes Distress Scale 2 is a 2 question prescreen that will be used to prescreen emotional burden. A score of 3 or higher on the DDS-2 will lead to the use of the 17-item survey.
Change in dietary intake for patients before and after delivery of the dietary intervention | three months
  The Dietary Screen Questionnaire (DSQ) will be administered to track changes in food habits before and after delivery of the intervention (session 2).
Beliefs about Medicines for patients and parent/caregiver over one year | 1 year
  Beliefs about Medicines Questionnaire (BMQ) is used to any change in patients beliefs and concerns about medications. It has been validated as a proxy for medication adherence.
Quality of life for patients | 1 year
  The Pediatric Quality of Life Inventory 3.2 (PedsQL 3.2) will be administered to assess changes in diabetes symptoms and management.

OTHER OUTCOMES:
Patient experience for patient and parent/caregiver | 1 year
  The Consumer Assessment of Healthcare Providers & Systems survey (CAHPS)assesses patient-clinician communication, experiences of discrimination based on race/ethnicity, insurance, and experiences leading to trust or distrust. Patient experience will be compared between control and intervention groups, both at baseline and at one year.
Demographic for Patients and Parents/Caregivers | baseline
  Self-reported demographic history (date of birth, gender, race and/or ethnicity, education, etc) will be collected.
Sociodemographic History for Parents/Caregivers | baseline
  Self-reported sociodemographic history (work status, marital members, household income, etc)
Implementation Outcome Measures for Research Staff | At end of study (end of 1 year)
  Implementation Outcome measure is used in behavioral health care as a psycho metric quality and will be used to assess how effectively clinic is being implemented.
Parent/Caregiver Clinic Satisfaction Survey | 1 year
  Survey will assess clinic satisfaction experience after each visit though a likert scale. Likert scale; "Strongly disagree" is 1, "disagree" is 2, "neutral" is 3, "agree" is 4, "strongly agree" is 5.
Shared Decision Making for Team Clinic Patients and Parents/Caregivers over one year | 1 year
  Shared decision making tool assess AYA and parent/caregiver's priorities for each medical visit using a mix of multiple choice and open-ended questions.
Research Team Appointment Satisfaction Survey | 1 year
  Survey will assess clinic satisfaction experience after each visit though a likert scale. Likert scale; "Strongly disagree" is 1, "disagree" is 2, "neutral" is 3, "agree" is 4, "strongly agree" is 5. Also, includes 4 open-ended questions to measures satisfaction for shared medical appointments.
Clinician Goals/Plans for Clinicians | 1 year
  Clinicians will work with families to discuss goals and plans guided by responding to 5 open-ended questions at each visit. Each member (Clinician, family, and AYA) will respond to these questions.
Healthcare Utilization Form | 1 year
  Healthcare Utilization Form is a 3-item survey that assess 911 call or emergency room usage for diabetic ketoacidosis, or severe hypoglycemia requiring glucagon.
Medication Review | baseline to one year
  General health history through review of participants EMR, completed by study coordinator
Adverse Events Form | baseline to one year
  The adverse events form will track any ED visits related to diabetes, DKA admissions, etc. throughout the study. It will be completed by Study Coordinator
Discontinuation and Termination Form | baseline to one year
  The discontinuation and termination form tracks reason for discontinuation of patient and agreement of continuation of medical records. To be completed by research coordinator.

CONTACTS AND LOCATIONS:
Overall Officials: Lily Chao, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No